CLINICAL TRIAL: NCT00452985
Title: Randomised Study With Docetaxel, Cisplatin and Cyclophosphamide vs Docetaxel and Carboplatin as First Line Chemotherapy With Advanced or Metastatic Ovarian Cancer
Brief Title: Docetaxel and Carboplatin as First-line Chemotherapy in Early Stage as Well as Advanced or Metastatic Ovarian Cancer
Acronym: OCSTUD
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: TAX_BD1_601
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: * Injection of Docetaxel
  * 3-hour gap
  * Injection of carboplatin
  Interventions: Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Docetaxel — 60-75 mg/m²
Drug: Carboplatin — AUC 5

SUMMARY:
Primary objective:

To assess response rate. To record the clinical improvement in relation to stage and histopathological grading.

Secondary objective:

To determine progression free survival. To find out overall survival. To evaluate the safety of the study regimen.

ELIGIBILITY:
Inclusion Criteria:

* Performance status Karnofsky index ≥ 60%.
* Early stage as well as advanced/metastatic ovarian cancer proven by abdominal ultrasonography, chest x-ray, Computerized axial tomography scan.
* Histologically: epithelial/germ cell
* Haematology: absolute neutrophil count: ≥2X10^9/L; Platelet: ≥150X10^9/L; Haemoglobin: ≥ 10g/dL
* Liver function: total bilirubin: ≤1X UNL (upper normal limit); Aspartate transaminase & Alanine aminotransferase: ≤2.5 x UNL; Alkaline phosphatase: ≤2.5 UNL
* Renal function: Creatinine: ≤130 µmol/L; If creatinine > 130 µmol/L, the 24 hour creatinine clearance should be > 60 ml/min.

Exclusion Criteria:

* Symptomatic peripheral neuropathy > grade 1 by National Cancer Institute - Common Toxicity Criteria scale
* Uncontrolled diabetes mellitus and uncontrolled hypertension
* Pregnant, or lactating patients(patients of childbearing potential must be using adequate contraception).
* Active infection or other serious underlying medical condition not compatible with program entry eg. congestive heart failure, previous myocardial infarction within 6 months prior to treatment.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 15 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced or metastatic ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2002-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Measurements of the disease (assessed clinically and/or by CA-125) | At baseline and from administration of drug to end of treatment
Response rate | From start to end of treatment
Clinical examination including neurologic examination, vital signs (blood pressure, heart rate, temperature), weight, assessment of any residual toxicity due to previous therapy, assessment of performance status. | From the beginning to the end of study
Adverse events | From the beginning to the end of the study

SECONDARY OUTCOMES:
Progression free survival | From administration of drug up to end of study
Overall survival | From administration of drug to end of study
Biology and Hematology laboratory determinations | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Rezaul-Farid Khan, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Dhaka, Bangladesh